CLINICAL TRIAL: NCT06415344
Title: A Long-term Extension Trial Investigating the Safety and Efficacy of GTX-102 in Patients With Angelman Syndrome
Brief Title: Long-term Extension of GTX-102 in Angelman Syndrome
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTX-102-CL302; 2024-510917-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GTX-102 (Experimental): Participants will receive GTX-102 via intrathecal lumbar puncture (IT LP) on a intrapatient flexible dosing schedule.
  Interventions: Drug: GTX-102

INTERVENTIONS:
Drug: GTX-102 — Antisense Oligonucleotide
  Other Names: apazunersen

SUMMARY:
The primary objective of the study is to evaluate the long-term safety profile of GTX-102 in participants with Angelman Syndrome (AS)

DETAILED DESCRIPTION:
This study is a phase 3, long term extension (LTE) which is open to participants rolling over from a prior GTX-102 clinical study. The LTE study will evaluate the long-term safety and efficacy of GTX-102 in participants with AS.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s).
* Completed a final study visit in a prior clinical trial with GTX-102. If the subject has an ongoing adverse event, medical monitor approval is required to rollover. The Screening visit must occur within 6 months of the last visit in the prior GTX-102 trial.
* From the time of informed consent through the end of the study and for at least 6 months after the final dose of GTX-102, females of childbearing potential who are sexually active must use highly effective contraception or abstinence. Males are able to participate if they agree to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the study and for at least 3 months after the final dose of GTX-102.

Exclusion Criteria:

* Discontinued from prior GTX-102 trial due to treatment-emergent adverse event assessed as related to GTX-102 and where the risk of study participation outweighs the benefits as deemed by the clinical judgment of the Investigator.
* History or evidence of any other medical, neurological, or psychological condition that would expose the subject to an undue risk of a significant AE or interfere with study assessments during the course of the trial as determined by the clinical judgment of the Investigator.
* Known hypersensitivity to GTX-102 or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects.
* Pregnant or breastfeeding or planning to become pregnant (self or partner) at any time during the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Frequency, Severity, and Relationship to Investigational Drug of Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | 5 Years

SECONDARY OUTCOMES:
Change from LTE Month 0 and Pretreatment in the Bayley-4 Raw Score | Month 0, 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceuticals Inc.
Locations (23):
- United States (6):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - University of California, San Diego - Rady Children's Hospital, San Diego, California
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
- Australia (2):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - The Royal Children's Hospital, Melbourne, Victoria
- Canada (5):
  - MAGIC Clinic Ltd, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Childrens Hospital London Health Sciences Centre, London, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
- France (2):
  - AP-HM - Hopital de la Timone, Marseille
  - AP-HP Hopital Necker-Enfants Malades, Paris
- Germany (2):
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
- Sheba Medical Center, Ramat Gan, Israel
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Sabadell
- United Kingdom (3):
  - University of Cambridge, Cambridge
  - Great Ormond Street Hospital for Children, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy Website — https://www.ultrarareadvocacy.com/conditions-we-study/angelman-syndrome-as/
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/
- See also: Ultragenyx Angelman Syndrome (AS) Research Study Opportunity — https://www.ultraclinicaltrials.com/angelman-syndrome-as/